CLINICAL TRIAL: NCT01456468
Title: Combination Therapy With Ursodeoxycholic Acid (UDCA) and All-Trans Retinoic Acid (ATRA) for Treatment of Primary Sclerosing Cholangitis - A Human Pilot Study
Brief Title: Combination Therapy With Ursodeoxycholic Acid (UDCA) and All-Trans Retinoic Acid (ATRA) for Treatment of Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James Boyer, Professor of Medicine, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012007734
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Cholangitis, Sclerosing
Keywords: Cholangitis, Sclerosing; Tretinoin; Ursodeoxycholic Acid
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UDCA + ATRA (Experimental): This is a single-arm study. All subjects will take UDCA and ATRA.
  Interventions: Drug: Oral all-trans retinoic acid (ATRA)

INTERVENTIONS:
Drug: Oral all-trans retinoic acid (ATRA) — The subjects will continue to take their current dose of UDCA (15 mg/kg/day), as per ongoing clinical care, and need to be on a stable dose of UDCA for at least six months prior to enrollment.
  The specific intervention is the addition of daily oral ATRA (45 mg/m^2) divided into 2 doses. To increase adherence to the dosing regimen, the drug will be compounded by the Research Pharmacies of Yale and Mayo into 2 formulations (30 mg and 40 mg capsules), and an Investigational New Drug (IND) permit was obtained for this process.
  Other Names: The medication is all-trans retinoic acid (ATRA).

SUMMARY:
The purpose of this research study is to determine whether the combination of UDCA and ATRA taken for 3 months will improve laboratory tests of liver and bile duct inflammation in patients with Primary Sclerosing Cholangitis (PSC). Our hypothesis is that a combination of these medications will improve the liver inflammatory tests in these patients, specifically a reduction in alkaline phosphatase (AP) by at least 30%.

DETAILED DESCRIPTION:
Patients with PSC often have ongoing inflammation and fibrosis (scars) along the length of their bile ducts, and eventually this involves the liver itself which can lead to cirrhosis (severe scarring), severe infections (cholangitis), bile duct cancer and death.

Although many patients are treated with UDCA, and experience improvement in their liver tests and relief of symptoms, no medical treatment to date has been found to produce a long-term improvement of inflammation and scarring, or to improved survival. For this reason, there is a great need to identify new medications which are effective for the treatment of PSC.

Recent work in animals by the research group at Yale University School of Medicine has shown that the combination of UDCA and ATRA produced a significant improvement in liver scarring and inflammation in animals with bile duct disease similar to that seen in PSC. This improvement included a lowering in the levels of bile acids, which are harmful to the liver, and a lowering of inflammation in the liver tissue of these animals. The benefits seen in this study were greater in animals receiving the combination of UDCA and ATRA compared to animals who received either medicine alone.

The medication ATRA is related to vitamin A, and has been used for many years as a topical medication in the treatment of skin conditions such as acne and psoriasis. It has also been used for nearly 20 years as an oral medicine in the treatment of a form of blood cancer (acute promyelocytic leukemia), where it is given for 90 days at a time. ATRA has been shown to produce a remission from the leukemia and is currently a standard treatment for patients with that specific condition. ATRA is not used routinely in the care of patients with liver or bile duct disease.

Based on the benefits observed by treatment with ATRA and UDCA in our animal studies, the investigators plan to study this combination in patients with PSC and believe that this may be an effective regimen for patients with this condition. The investigators will check blood tests of the liver and bile ducts before, during, and after the treatment in order to look for changes to liver tests which would be due to the medication combination.

Therefore, the goal of this study is to study the changes to liver tests in patients with PSC who take a combination of UDCA and ATRA for 90 days, comparing levels at the beginning of the study to those at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PSC for at least 6 months, made by clinical evaluation in addition to one of the following: a prior endoscopic retrograde cholangiography (ERC), magnetic resonance cholangiography (MRC, also termed MRI/MRCP) or liver biopsy.
* Progressing disease or stable disease with persistent elevation in AP despite treatment with UDCA (15 mg/kg/day) for at least 6 months.

  * Measures of progressing disease:

    1. Cholangitis within the past 12 months.
    2. Presence or progression of biliary abnormalities on MRI/MRC.
    3. Elevated liver tests (alkaline phosphatase, bilirubin, aspartate aminotransferase [AST], alanine aminotransferase [ALT]).
* Age between 18 and 80.

Exclusion Criteria:

* Pregnancy or planned pregnancy during study period and within 6 months of study completion.
* Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher cardiac disease, hyperlipidemia, hypertriglyceridemia, hepatic injury, or adverse event related to administration of UDCA or ATRA.
* Prior intolerance to UDCA or ATRA (or related oral vitamin A compounds).
* Evidence of decompensated cirrhosis within the past 6 months (i.e. variceal bleeding, uncontrolled ascites, hepatic encephalopathy, jaundice).
* Estimated need for liver transplantation within 1 year.
* Any evidence of hepatocellular carcinoma, cholangiocarcinoma, or other malignancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement in serum alkaline phosphatase levels | Baseline and after 3 months of treatment.
  The primary outcome measure is a 30% improvement in serum alkaline phosphatase in subjects, comparing pre- and post-treatment values for each individual.

CONTACTS AND LOCATIONS:
Overall Officials: James L Boyer, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University School of Medicine - 333 Cedar St - 1080 LMP, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] He H, Mennone A, Boyer JL, Cai SY. Combination of retinoic acid and ursodeoxycholic acid attenuates liver injury in bile duct-ligated rats and human hepatic cells. Hepatology. 2011 Feb;53(2):548-57. doi: 10.1002/hep.24047. Epub 2010 Dec 10. PMID 21274875